CLINICAL TRIAL: NCT06645327
Title: Utility of the Superior Vena Cava Collapsibility Index (SVC-CI) to Predict Fluid Responsiveness in Patients With Coronary Artery Disease Undergoing Surgical Revascularization
Acronym: SVC-CI
Status: Recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Edward Stredny, MD, Assistant Professor, Department of Anesthesiology and Perioperative Medicine, Penn State Health Milton S Hershey Medical Center
Other Study IDs: STUDY 24328; Study 24328 (Other: Penn State Health Penn State Hershey Medical Center)
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Bypass Grafting Surgery (CABG)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: (LVEF>40%)
  Interventions: Other: a change in operating room table position, which will mimic an IV fluid bolus
- Group 2: (LVEF<40%),
  Interventions: Other: a change in operating room table position, which will mimic an IV fluid bolus

INTERVENTIONS:
Other: a change in operating room table position, which will mimic an IV fluid bolus — Cardiac Output (CO) measurements will be obtained at two separate time points: prior to sternotomy (opening of the chest) and after separation from cardiopulmonary bypass.
  Intervention
  1. the participant will be placed in the reverse Trendelenburg position (head up) to 15 degrees for 60-90 seconds. CO measurement will be obtained
  2. the participant will be transitioned to the Trendelenburg position (head down) to 15 degrees for 60-90 seconds. CO measurement will be obtained

SUMMARY:
To investigate the superior vena cava collapsibility index (SVC-CI), measured via transesophageal echocardiography (TEE), as a marker of fluid responsiveness. Two groups will be compared in this study. Groups will be identified by obtaining cardiac output (CO) by standard means using the TEE or pulmonary arterial catheter (PAC). Both of these monitors are considered standard for patient's undergoing coronary artery bypass grafting surgery (CABG) and recording initial CO readings. Based on CO, the patient's will be placed in study groups one or two. Participants with normal and mildly reduced left ventricular ejection fraction (LVEF >40%) for group one and those with moderately to severely reduced LVEF (<40%) in the second group.

Following group separation, we will measure the SVC-CI and CO metric in both groups. The intervention will be an operating room table tilt test (head up and then head down) to artificially simulate giving the patient additional fluid. Before and after table tilt, the SVC-CI and CO will be obtained and measured. The SVC-CI is a mathematical equation determined by distance measurements taken via TEE to identify how much the superior vena cava has collapsed following table tilt. Participants will be considered responders if the CO increases by 12% following intervention. Non responders less than 12% change in CO following intervention. Our hypothesis is that the SVC-CI can differentiate responders vs non-responders with regards to fluid responsiveness with adequate sensitivity and specificity in participants with CAD undergoing isolated CABG. The SVC-CI numerical values for the two groups, responders and non-responders, will calculate a threshold of sensitivity and specificity percentages for future patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Participants with CAD undergoing CABG utilizing cardiopulmonary bypass
3. Participants who are able to consent for themselves
4. Primary language is English

Exclusion Criteria:

1. Age less than 18 years of age
2. Participants with CAD undergoing off-pump coronary artery bypass (OP-CAB)
3. Severe cardiac valvular pathologies or active congestive heart failure
4. Participants in active arrhythmia such as atrial fibrillation and atrial flutter at the time of data collection.
5. Participants who are unable to consent for themselves
6. Primary language is something other than English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CAD undergoing CABG utilizing cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To determine an appropriate cut-off value for the SVC-CI in participants with CAD undergoing isolated CABG to distinguish volume responders from non-responders. | 10 minutes of time added to your surgery time.
  1. Responders increases by 12% or more following intervention
  2. Non responders less than 12% change in CO following intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
It will depend if the data is shared in data bases and what kind of data bases. this has not been determined.

REFERENCES:
- [Background] 1. Charbonneau H, Riu B, Faron M, et al. Predicting preload responsiveness using simultaneous recordings of inferior and superior vena cavae diameters. Crit Care. 2014;18(5):473. 2. Hrishi AP, Sethuraman M, Menon G. Quest for the holy grail: Assessment of echo-derived dynamic parameters as predictors of fluid responsiveness in patients with acute aneurysmal subarachnoid hemorrhage. Ann Card Anaesth. 2018;21(3):243-248. 3. Vieillard-Baron A, Chergui K, Rabiller A, et al. Superior vena caval collapsibility as a gauge of volume status in ventilated septic patients. Intensive Care Med. 2004;30(9):1734-1739. 4. Vignon P, Repessé X, Bégot E, et al. Comparison of Echocardiographic Indices Used to Predict Fluid Responsiveness in Ventilated Patients. Am J Respir Crit Care Med. 2017;195(8):1022-1032.